CLINICAL TRIAL: NCT00057213
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Flexible-Dose Study Evaluating Efficacy, Safety, and Tolerability of Once-Daily Oral GW353162 (20-40-60mg) Versus Placebo in Subjects With Major Depressive Disorder Over an Eight-Week Treatment Period.
Brief Title: An 8 Week Study Of Depression In Adults Diagnosed With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHB20002
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder (MDD),; Flexible; GW353162,
MeSH Terms: conditions — Depressive Disorder, Major | interventions — radafaxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Radafaxine

SUMMARY:
A Placebo Controlled Study Evaluating Efficacy, Safety and Tolerability of Medication in Patients with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD)
* Duration of current depressive episode 12 weeks - 24 months
* Patients can read and write at a level sufficient to provide a signed consent
* If female, patients must be practicing an acceptable method of birth control

Exclusion Criteria:

* Patients have other psychiatric disorders that would affect patient's response to treatment
* Patients have not responded to two or more adequate courses of antidepressant therapy
* Patients cannot be currently abusing illicit drugs or alcohol
* Patients are not currently receiving psychotherapy
* Patients have received electroconvulsive therapy within 6 months prior to screening
* Patients are pregnant or lactating

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 367 (Actual)
Dates: Start 2003-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) after 8 weeks of treatment | 8 Weeks

SECONDARY OUTCOMES:
Change in the MADRS score at other timepoints; change in Clinical Global Impression; percentage of remitters and responders based on the MADRS; change in disability, motivation, energy, fatigue and pain;incidence of adverse events over course of study;

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Florence, Kentucky
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Lyndhurst, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Salt Lake City, Utah